CLINICAL TRIAL: NCT07405957
Title: Effects of Naturally Occurring Lions Mane Extract on Cognitive Performance, Serum Biomarkers and Indices of Affect (Pro00083830)
Brief Title: Effects of Two Different Lion's Mane Extracts (Lions Mane Fruiting Body & Lions Mane Fruiting Body With Mycellium) on Cognitive Performance, Subjective Affect, Serum Biomarkers, and Gut Microbiota in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Food Sciences Inc. (Industry)
Collaborators: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AFS-01-2024
Record Dates: First submitted 2026-01-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult Females; Healthy Adult Male
Keywords: Randomized, double blind, placebo controlled, Lions Mane; Hericium erinaceus; Fruiting Body; Mycelium
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nordic Lions Mane (Hericium erinaceus) fruiting body extract (Experimental): 1 gram / day of active lions mane or placebo
  Interventions: Dietary Supplement: Lions Mane (Hericium erinaceus) Fruiting body and mycelium
- Lions Mane (Hericium erinaceus) fruiting body and mycelium extract (Active Comparator): Lions Mane (Hericium erinaceus) fruiting body and mycelium extract combined in equal portions
  Interventions: Dietary Supplement: Lion Mane (Hericium erinaceus) fruiting body extract - Nordic Origin
- Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Other: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Lion Mane (Hericium erinaceus) fruiting body extract - Nordic Origin — This extract contains only fruiting body of the Hericium erinaceus
  Arms: Lions Mane (Hericium erinaceus) fruiting body and mycelium extract
Dietary Supplement: Lions Mane (Hericium erinaceus) Fruiting body and mycelium — This extract contains both the fruiting body and the mycelium of the Hericium erinaceus, providing different levels of active triterpenoids and beta glucans than fruiting body alone.
  Arms: Nordic Lions Mane (Hericium erinaceus) fruiting body extract
Other: Maltodextrin (Placebo) — Maltodextrin (Placebo)
  Arms: Maltodextrin

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel-arm study design, of healthy men and women assigned to one of three groups: 1 gram/day of MycothriveTM Nordic origin fruiting body lion's mane (M-LM), 1 gram/day of a commercially available mycelium and fruiting body lion's mane (MFB-LM), or placebo (PL) to evaluate Lions mane potential cognitive and gut health benefits in a controlled daily dose for 45 days.

DETAILED DESCRIPTION:
Lion's Mane (LM) contains β-glucan polysaccharides, proteins, polyketides, hericenones and erinacine terpenoids, cyathane diterpenoids, lectins, phenols, isoindolinones, sterols, and myconutrients, which have been found to provide cognitive and neuroprotective properties. Erinacines within the mycelium of lions mane have demonstrated nootropic effects through the stimulation of nerve growth factor (NGF) synthesis, which plays a critical role in the growth, maintenance, and survival of neurons within the central nervous system, particularly the basal forebrain cholinergic system. Acute affects were shown to improve working memory, complex attention, and reaction time and perceptions of happiness in Lions Mane Fruiting body. This study aims to determine key differences (if any) in cognitive tasks, subjective affect (e.g., VAS scales for mental clarity, memory, mood, focus, concentration), serum biomarkers (BDNF, TNF-alpha,IL-6, HS-CRP), microbiome (alpha & beta diversity, keystone species, etc.) with daily consumption.

ELIGIBILITY:
Inclusion Criteria: Provide voluntary signed and dated informed consent.

* Be in good health and able to participate in cognitive performance testing as determined by assessment, medical history, and routine blood chemistries.
* Between the of 40 and 65 years of age (inclusive).
* Body Mass Index of 18.5-39.9 (inclusive).
* Body weight of at least 110 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5-minute) rest period, and two more measurements will be taken.

The average of all three measurements will be used to determine eligibility.

* Normal supine, resting heart rate (<90 per minute).
* Able to provide an adequate blood draw.
* If a dietary supplement was initiated within the past month, the participant is willing to discontinue supplement use followed by a 2-week washout prior to participation in the study.
* Willing to duplicate their previous 24-hour diet, refrain from caffeine for 12 hours, refrain from exercise for 24 hours prior to each trial, and fast for 8 hours prior to each visit.

Exclusion Criteria:Smokes more than 10 cigarettes per day or uses other nicotine products (i.e. vape, patch) that deliver a similar amount of nicotine.

* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. electrolyte abnormalities, diabetes, thyroid disease, adrenal disease, hypogonadism, short bowel syndrome, diarrheal illnesses, history of colon resection, gastric ulcer, reflux disease, gastroparesis, Inborn-Errors-of-Metabolism (such as PKU). Chronic medically diagnosed inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Medical history of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Medical history of a cognitive or psychiatric disorder.
* Currently using medications to treat anxiety or depression.
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates- of-Analysis.
* Women currently pregnant, trying to become pregnant or breastfeeding a child.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Cognitive function measured by Composite memory (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome composite memory (Unit of Measure = milliseconds)
Cognitive Performance in visual memory, Unit of Measure = milliseconds | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome visual memory, Unit of Measure = milliseconds
Cognitive Function in verbal memory (the ability to recognize, remember, and retrieve words and geometric figures). (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome Measure verbal memory (the ability to recognize, remember, and retrieve words and geometric figures). (Unit of Measure = milliseconds)
Cognitive Function in reaction time (the ability to react to a simple and increasingly complex direction set) (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome measure: reaction time (the ability to react to a simple and increasingly complex direction set) (Unit of Measure = milliseconds)
Cognitive flexibility (the ability to adapt to rapidly changing and increasingly complex set of directions) (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome measure: cognitive flexibility (the ability to adapt to rapidly changing and increasingly complex set of directions) (Unit of Measure = milliseconds)
Cognitive Function measured by executive function (the ability to recognize rules and categories, and manage or navigate rapid decision making) (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome Measure: executive function (the ability to recognize rules and categories, and manage or navigate rapid decision making) (Unit of Measure = milliseconds)
Cognitive Function measured by motor speed (the ability to perform movements to produce and satisfy an intention towards a manual action and goal) (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome Measure: motor speed (the ability to perform movements to produce and satisfy an intention towards a manual action and goal) (Unit of Measure = milliseconds)
Cognitive Function measured by psychomotor speed (the ability to perceive and respond to visual-perceptual information and perform motor speed and fine motor coordination) (Unit of Measure = milliseconds) | 45 days
  Cognitive performance will be assessed using CNS Vital Signs, a computerized neurocognitive testing platform that provides a validated assessment of cognitive function. Outcome Measure: psychomotor speed (the ability to perceive and respond to visual-perceptual information and perform motor speed and fine motor coordination) (Unit of Measure = milliseconds)

SECONDARY OUTCOMES:
Microbiome Diversity namely Faecalibacterium prausnitzii (expressed as copies per gram stool). | 45 days
  Between and within-group changes in microbiome (alpha & beta diversity, keystone species, namely Faecalibacterium prausnitzii expressed as copies per gram stool). (Diagnostic Solutions Laboratory Alpharetta, GA).

OTHER OUTCOMES:
Heart rate measured in BPM | 45 days
  Safety heart rate (BPM)
Blood Presure measured by Systolic BP (mm Hg) Diastolic BP (mm Hg) | 45 Days
  Description: Safety blood pressure: Systolic BP (mm Hg) Diastolic BP (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. La Monica, Ph.D., CSCS, Principal Investigator — The Center for Applied Health Sciences
Locations (1):
- Center for Applied Health Sciences, Canfield, Ohio, United States